CLINICAL TRIAL: NCT06773065
Title: The Role Of Central Sensitisation In Women With Endometriosis: A Prospective Observational Study
Brief Title: Central Awareness in Women With Endometriosis
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: STUDIO CS 2021
Record Dates: First submitted 2024-12-01; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Endometriosis
Keywords: endometriosis; central awareness; central sensitisation syndrome
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gathering some information obtained during the gynaecological examination and transvaginal ultrasound check-up to be able to assess the prevalence of Central Sensitisation Syndrome (CSS) in women with endometriosis and also to be able to assess related risk factors. CSS has been defined as an algic syndrome due to a hyperactivation of the sensitivity circuit at a central level; the diagnosis is based on the result obtained from a questionnaire, the Central Sensitisation Inventory (CSI), which evaluates the presence and intensity of 25 clinical symptoms. For this reason, a questionnaire is proposed to be completed at the time of the check-up visit.

DETAILED DESCRIPTION:
Endometriosis is a chronic benign condition characterised by the presence of endometrial cells within the uterine wall and/or in anatomical locations outside the uterus; 1 in 10 women of reproductive age are affected. Various symptoms are associated with endometriosis: dysmenorrhoea, chronic pelvic pain, peri-ovulatory pain, dyspareunia, dyschezia, dysuria. Chronic pelvic pain (CPD) is one of the most common symptoms of clinical manifestation of endometriosis; 71% to 87% of women surgically diagnosed with endometriosis suffer from it. Therapies have focused on hormone therapy and surgery; although they can control the extent of the disease, most patients fail to resolve DPC. It has therefore been suggested to consider a polycentric chronic pelvic pain (DPC) origin perspective, as suggested by the myofascial and central sensitisation syndrome, which seem to contribute to pain through activation of different trigger points.

In central sensitisation (CS), peripheral nociceptive signal transmission pathways (such as those due to the presence of endometriosis lesions) can lead to adaptive changes in neurons of the central nervous system, including presynaptic effects (e.g. changes in neurotransmitter release) and postsynaptic effects (e.g. increased calcium entry into N-methyl-D-aspartate channels). This leads to a reduction in the activation threshold of central neurons and consequently to a hypersensitisation to pain associated with symptoms of hyperalgesia and allodynia. Together with pain, other symptoms of central sensitisation may occur, such as fatigue, depression, hypersensitivity. While the direct innervation of endometriotic lesions results in the activation of visceral nociception and peripheral sensitisation, CS creates a pain-feeding circuit that is independent of the underlying pathology. In some women with endometriosis, hyperalgesia, allodynia, psychological comorbidities and extension of receptor zones have been observed. Neuroimaging studies have identified changes in the grey matter in women with endometriosis and chronic pelvic pain, further supporting the hypothesis of a central component in women with endometriosis.

CS in some pathologies has led to the definition of a true algic syndrome, called Central Sensitisation Syndrome (CSS). For the identification of this syndrome in clinical practice, the Central Sensitisation Inventory (CSI) has been proposed. It takes the form of a screening tool, based on the patient's completion of a questionnaire, and helps to determine the severity of the symptoms characteristic of this syndrome, enabling its diagnosis. The CSI has been studied and validated for the diagnosis of CSS in patients suffering from fibromyalgia, irritable bowel syndrome and migraine.

Despite the practicality and applicability of the CSI, there appears to be only one study in the literature evaluating its application in women with endometriosis. In particular, this study analyses the correlation between the CSI score and two symptoms characteristic of endometriosis: deep dyspareunia and bladder and/or pelvic floor pain. To date, there appear to be no studies in the literature reporting the prevalence of CSS in patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Women with a clinical, ultrasound and/or surgical diagnosis of endometriosis
* Aged between 18 and 50 years
* Patients starting or already taking hormone therapy
* Patients coming for a first visit or outpatient follow-up visit
* Signature of informed consent to participate in the study

Exclusion Criteria:

* Post-menopausal women (spontaneous or iatrogenic)
* Virgo patients
* Patients with poor compliance with hormone therapy, who are not taking it properly or have discontinued therapy spontaneously
* Positive history of any malignant neoplasm
* Positive medical history of specific medical conditions that adversely affect the central nervous system, such as: brain or spinal cord damage, neurological diseases or peripheral nerve damage, multiple sclerosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of central sensitisation syndrome (CSS) | At the first visit after enrollment
  Prevalence of CSS in women with endometriosis by Central Sensitization Inventory (CSI) questionnaire. It consists of two parts:
  * A: assesses clinical symptoms related to CSS, based on the frequency of each symptom, with a subjective scale from 0 (never) to 4 (always), the maximum score is 100. Higher scores are associated with a higher degree of symptomatology reported by the patient.
  * B: previous diagnosis of restless legs syndrome, chronic fatigue syndrome, fibromyalgia, temporomandibular disorders, migraine or headache, irritable bowel syndrome, multiple chemical sensitivity cervical lesions, anxiety or panic attacks, depression. 7 are typical of CSS if 3 are closely related to CSS. Patients are asked whether they have ever been diagnosed with one of the conditions and in which year they were diagnosed.
  The total score on Part A will then be calculated and the presence or absence o of CSS diagnoses noted.
  CSS will be defined as a score greater than or equal to 40.

SECONDARY OUTCOMES:
Difference in mean value of the Central Sensitization Inventory (CSI) score | At the first visit after enrollment
  Difference in mean value of the CSI score in women with endometriosis in relation to response to hormone therapy.
  It consists of two parts:
  * A: assesses clinical symptoms related to CSS, based on the frequency of each symptom, with a subjective scale from 0 (never) to 4 (always), the maximum score is 100. Higher scores are associated with a higher degree of symptomatology reported by the patient.
  * B: previous diagnosis of restless legs syndrome, chronic fatigue syndrome, fibromyalgia, temporomandibular disorders, migraine or headache, irritable bowel syndrome, multiple chemical sensitivity cervical lesions, anxiety or panic attacks, depression. 7 are typical of CSS if 3 are closely related to CSS. Patients are asked whether they have ever been diagnosed with one of the conditions and in which year they were diagnosed.
  The total score on Part A will then be calculated and the presence or absence o of CSS diagnoses noted. CSS will be defined as a score greater than or equal to 40
Correlation of the CSI value with the degree of various endometriosis symptoms | At the first visit after enrollment
  Correlation of the CSI value with the degree of various endometriosis symptoms assessed on a Visual Analogue Scale (VAS) from 0 (no pain) to 10 (worst pain)
Correlation of the CSI value with the time duration of hormone therapy | At the first visit after enrollment
  Correlation of the CSI value with the time duration of hormone therapy
Correlation of the CSI value with the localizazion of endometriosis lesions | At the first visit after enrollment
  Correlation of the CSI value with the localization of endometriosis lesions
Correlation of the CSI value with other clinical characteristics | At the first visit after enrollment
  Correlation of the CSI value with other clinical characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Diego Raimondo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy